CLINICAL TRIAL: NCT05600218
Title: Real World Andalusian Multicenter Data on Patients With Pulmonary Arterial Hypertension Treated With IP Prostacyclin Receptor Agonists
Brief Title: RWD Patients With Pulmonary Arterial Hypertension Treated With IP Prostacyclin Receptor Agonists
Acronym: RAMPHA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Costa del Sol (Other)
Collaborators: Hospital Universitario Virgen Macarena (Other); Hospital Regional de Malaga (Other); Hospital Universitario Virgen de la Victoria (Other); Hospital San Juan de la Cruz (Other); Complejo Hospitalario de Especialidades Juan Ramón Jimenez (Other); Hospitales Universitarios Virgen del Rocío (Other); Hospital Clinico Universitario San Cecilio (Other); Hospital Universitario de Valme (Other); Hospital de Poniente (Unknown)
Responsible Party: Principal Investigator, Rafael Bravo Marqués, Medical Specialist, Department of Cardiology, Hospital Costa del Sol, Marbella (Malaga,) Spain, Hospital Costa del Sol
Other Study IDs: 0991-N-21
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Selexipag; Real World Data; Effectiveness
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Cohort 1: Patients with pulmonary arterial hypertension on treatment with prostacyclin IP receptor agonists because they are at intermediate risk of mortality at one year
  Interventions: Drug: No intervention - Observational study

INTERVENTIONS:
Drug: No intervention - Observational study — Real life drug evaluation

SUMMARY:
This is an observational, ambrispective study of patients in real world clinical practice, who has pulmonary arterial hypertension in whom a prostacyclin IP receptor agonist (Selexipag) is initiated between 2017 and 2021.

The aim of this study answer the following questions:

* Changes in the mortality risk profile of these patients after treatment administration.
* Baseline characteristics of patients initiating Selexipag.
* Parameters used for risk stratification prior to treatment escalation.
* Events during follow-up.

No comparison group available

ELIGIBILITY:
Inclusion Criteria:

* They agree to participate in the study by signing an informed consent form

Exclusion Criteria:

* Decline to participate in the study
* Patients living 6 months or less in the reference health area
* Patients with active malignant tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary arterial hypertension (mostly intermediate risk patients) who are started on treatment with Selexipag according to clinical practice guideline recommendations.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement (risk profile) | 12 months
  Percentage of patients reducing annual mortality risk profile according to ESC/ERS Clinical Practice Guidelines 2015 Risk Stratification.

SECONDARY OUTCOMES:
Risk stratification variables | Basaline
  Percentage of clinical tests that have been used to include study treatment.
Events | 12 months
  Incidence of events in follow-up: admission for worsening pulmonary hypertension; need for systemic prostacyclins; unscheduled admission for any cause; death related to pulmonary hypertension; death from any cause.

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Hospital de Poniente, El Ejido, Almería
  - Hospital San Juan de la Cruz, Úbeda, Jaén
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Clinico Universitario San Cecilio, Granada
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital Regional de Malaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Valme, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Undecided
Once the database has been completed and the main results article has been published, access to the database through a free repository (e.g. Mendeley) will be considered.